CLINICAL TRIAL: NCT03584724
Title: Assessment of the Anti-inflammatory Effects of Norflo Oro in Acute Relapses of HLA-B27 Associated Autoimmune Uveitis: a Multicenter Randomized, Placebo Controlled, Double-blind Clinical Study
Brief Title: Assessment of the Anti-inflammatory Effects of Norflo Oro in Acute Relapses of HLA-B27 Associated Autoimmune Uveitis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Eye Pharma (Industry)
Collaborators: Bascom Palmer Eye Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Norflo-Oro-16
Record Dates: First submitted 2018-04-26; First posted 2018-07-12 (Actual); Results first posted 2022-03-28 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Uveitis
Keywords: HLA-B27; relapses; curcumin
MeSH Terms: conditions — Uveitis; Recurrence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Up to 60 eligible patients will be randomly assigned to NORFLO® ORO or placebo treatment groups in a 1:1 ratio using a stratified randomization blocks scheme.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Norflo Oro (Experimental): The study subject will take the entire content of one packet of Norflo (each box contains 30 packets) with meal twice per day for one year. The study subject will be evaluated in a total of three visits.
  Interventions: Drug: Norflo Oro
- Placebo for Norflo Oro (Placebo Comparator): The study subject will take the entire content of one packet of Placebo (each box contains 30 packets) with meal twice per day for one year. The study subject will be evaluated in a total of three visits.
  Interventions: Drug: Placebo for Norflo Oro

INTERVENTIONS:
Drug: Norflo Oro — Norflo Oro is highly bioavailable curcumin complexed into phytosomes
  Other Names: Meriva
  Arms: Norflo Oro
Drug: Placebo for Norflo Oro — Placebo consist of look-alike single foil pouches without active ingredient of Norflo.
  Other Names: Placebo
  Arms: Placebo for Norflo Oro

SUMMARY:
The purpose of this study is to explore the efficacy of Norflo Oro in the treatment of relapsing autoimmune uveitis (RAU), measured as a long term reduction of the frequency and the severity of relapses, in patients with HLA-B27 associated uveitis, under conditions of routine medical practice. The reduction of the mean number of relapses per patient between the year before study treatment and the study period will also be assessed.

DETAILED DESCRIPTION:
The secondary objective of this study will be: (i) evaluation of the improvement of side effects due to HLA-B27 associated uveitis such as intraocular pressure (IOP), cystoid macular edema, keratophaty and synechia (ii) evaluation of the improvement in uveitis-related symptoms: BCVA and symptoms measured by VAS, like ocular pain, photophobia, floaters and blurred vision; (iii) evaluation of cell damage and inflammation reduction in patients with HLA-B27 associated uveitis; (iv) evaluation of the patients' attitude towards the study treatment and also the evaluation of the safety profile of the study product.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of HLA-B27 positive related uveitis in non- acute phase
* At least one autoimmune uveitis relapse

Exclusion Criteria:

* Use of supplements (nutraceuticals) or systemic therapy for uveitis with anti-inflammatory immunosuppressive or biological drugs within last 30 days
* Anticipated need for systemic anti-inflammatory treatment during the study
* Use of intravitreal peribulbar, sub-tenon, periocular injection in the previous 6 months
* Long-term treatment with a systemic anti-inflammatory, immune suppressant drugs
* Woman taking hormonal contraceptives, pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2020-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pia Allegri, Principal Investigator — S.S. Uveitis Center, Rapallo Hospital, Genoa- Italy
Locations (1):
- Bascom Palmer Eye Institute, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allegri P, Mastromarino A, Neri P. Management of chronic anterior uveitis relapses: efficacy of oral phospholipidic curcumin treatment. Long-term follow-up. Clin Ophthalmol. 2010 Oct 21;4:1201-6. doi: 10.2147/OPTH.S13271. PMID 21060672
- [Background] Steigerwalt R, Nebbioso M, Appendino G, Belcaro G, Ciammaichella G, Cornelli U, Luzzi R, Togni S, Dugall M, Cesarone MR, Ippolito E, Errichi BM, Ledda A, Hosoi M, Corsi M. Meriva(R), a lecithinized curcumin delivery system, in diabetic microangiopathy and retinopathy. Panminerva Med. 2012 Dec;54(1 Suppl 4):11-6. PMID 23241930
- [Background] Mazzolani F, Togni S. Oral administration of a curcumin-phospholipid delivery system for the treatment of central serous chorioretinopathy: a 12-month follow-up study. Clin Ophthalmol. 2013;7:939-45. doi: 10.2147/OPTH.S45820. Epub 2013 May 22. PMID 23723686
- [Derived] Allegri P, Cimino L, Davis JL, Tugal-Tutkun I; Norflo Oro study group. Assessment of the Anti-inflammatory Effects of NORFLO(R) ORO in Acute Relapses of HLA-B27-associated Autoimmune Uveitis: A Multicenter, Randomized, Placebo-controlled, Double-blind Clinical Study. Ocul Immunol Inflamm. 2023 Apr;31(3):526-535. doi: 10.1080/09273948.2022.2039210. Epub 2022 Mar 30. PMID 35353651

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Norflo Oro | Placebo for Norflo Oro
Started | 25 | 24
Completed | 18 | 23
Not Completed | 7 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Norflo Oro | Placebo for Norflo Oro | Total
Number analyzed (Participants) | 25 | 24 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 19 | 41
  >=65 years | 3 | 5 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.40 (13.21) | 50.88 (14.90) | 48.59 (14.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 13 | 13 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 23 | 23 | 46
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 25 | 23 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 5
  Italy | 19 | 19 | 38
  Turkey | 3 | 3 | 6
Relapses Per Patient [Mean (Standard Deviation); unit: Relapses] — Number of relapses as episodes of uveitis recurrence
  Relapses | 1.95 (0.94) | 1.50 (0.83) | 1.71 (0.94)

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Number of Uveitis Relapses Per Patient Between the 12 Month Study Period Compared to Baseline
Description: The mean number of uveitis relapses per patient in the 12 months of study duration (12 months) will be compared to the average number of uveitis relapses per patient in the 12 months before (baseline) for the Norflo Oro group and for the Placebo group.
Time Frame: Baseline and 12 months
Population: Only patients that completed the 12 month study were included in the analysis of the mean number of relapses per patient during the study duration (12 months).
Measure: Mean (Standard Deviation); unit: Relapses Per Patient
Arm/Group | Norflo Oro | Placebo for Norflo Oro
Number analyzed (Participants) | 20 | 24
Relapses Per Patient | 0.35 (0.75) | 0.58 (0.88)

2. Secondary Outcome: Changes in Side Effects Associated With HLA-B27 Uveitis
Description: The changes in side effects associated with HLA-B27 uveitis, such as intraocular pressure (IOP) in the NORFLO® ORO treatment group and control group at the end of the study (12 month) compared to the 12 months before the study started (baseline)
Time Frame: 12 months
Population: Only participants that completed the study were included in the 12-month evaluation
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Norflo Oro | Placebo for Norflo Oro
Number analyzed (Participants) | 20 | 24
mmHg
  IOP change (right eye) | 0.44 (1.85) | 0.22 (3.01)
  IOP change (left eye) | -0.06 (1.70) | -0.09 (2.37)

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse Events were monitored/assessed without regard to the specific Adverse Event Term.
Arm/Group | Norflo Oro | Placebo for Norflo Oro
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/24
Serious Adverse Events (participants affected / at risk) | 3/20 | 0/24
Other Adverse Events (participants affected / at risk) | 20/20 | 19/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Norflo Oro (N=20) | Placebo for Norflo Oro (N=24)
wrist fracture (Musculoskeletal and connective tissue disorders) | 1 | NA
drink poisoning (Injury, poisoning and procedural complications) | 1 | NA
Fracture of the foot (Musculoskeletal and connective tissue disorders) | 1 | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Norflo Oro (N=20) | Placebo for Norflo Oro (N=24)
eye disorders (Eye disorders) | 4 (16) | 7 (13)
gastrointestinal disorders (Gastrointestinal disorders) | 12 (34) | 10 (18)
General disorders and administration site conditions (General disorders) | 4 (4) | 3 (4)
Infections and infestations (Infections and infestations) | 8 (16) | 8 (14)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 4 (4) | 2 (3)
investigations (Investigations) | 0 (0) | 1 (1)
metabolism and nutrition disorders (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Muskoloskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 2 (5) | 5 (9)
nervous system disorders (Nervous system disorders) | 5 (22) | 7 (10)
renal and urinary disorders (Renal and urinary disorders) | 2 (2) | 0 (0)
respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
vascular disorders (Vascular disorders) | 2 (2) | 3 (3)
ear and labyrinth disorders (Ear and labyrinth disorders) | 0 (0) | 1 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-10-10): https://cdn.clinicaltrials.gov/large-docs/24/NCT03584724/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-20): https://cdn.clinicaltrials.gov/large-docs/24/NCT03584724/SAP_001.pdf